CLINICAL TRIAL: NCT03026088
Title: A Single-arm, Interventional, Multi-center, Pilot Study to Evaluate the Efficacy of Oral Bisoprolol on Heart Rate Reduction in Chinese Chronic Heart Failure Patients With NYHA Class II - IV (Biso-CHF Study)
Brief Title: Efficacy of Oral Bisoprolol on Heart Rate Reduction in Chinese Chronic Heart Failure Participants
Acronym: Biso-CHF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited beta-blocker naive participants among newly diagnosed heart failure participants, which led barrier to the recruitments.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Co., Ltd., China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS200006-0039
Record Dates: First submitted 2017-01-12; First posted 2017-01-20 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Heart Failure
Keywords: Chronic Heart Failure; Bisoprolol; Heart rate control
MeSH Terms: conditions — Heart Failure | interventions — Bisoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bisoprolol (Experimental)
  Interventions: Drug: Bisoprolol

INTERVENTIONS:
Drug: Bisoprolol — Participants received Bisoprolol orally, once daily at a dose of 1.25 milligram (mg) up to Weeks 3, and then it was up-titrated to 2.5 mg up to Week 6, 3.75 mg up to Week 10, 5 mg up to Week 14, 7.5 mg up to Week 18 and 10 mg up to Week 26.
  Other Names: Brand name: Concor

SUMMARY:
This is a single-arm, open label, interventional, multi-center, phase 4 pilot study.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 year, male or female.
* Chronic Heart failure subjects with medical history of cardiac disease or other related cardiovascular disease.
* Left ventricular ejection fraction (LVEF) less than or equal to (=<) 40 percent (%).
* New York Heart Association (NYHA) class of II - IV
* NYHA II ： Slight limitation of physical activity. Comfortable at rest, but ordinary physical activity results in undue breathlessness, fatigue or palpitation.
* NYHA III：Marked limitation of physical activity. Comfortable at rest, but less than ordinary activity causes undue breathlessness, fatigue or palpitation.
* NYHA IV：Unable to carry on any physical activity without discomfort. Symptoms at rest can be present. If any physical activity is undertaken, discomfort increased.
* Signed Informed Consent Form (ICF).

Exclusion Criteria:

* Acute coronary syndrome (ACS) within 3 months.
* Under beta-blocker treatment for the last 2 weeks.
* Under other medicine treatment which may affect heart rate, like Non-dihydropyridine calcium channel blockers (NDHP-CCBs) or ivabradine for the last 2 weeks; Under Digoxin treatment [more than (>) 0.125 milligram (mg)].
* Uncontrolled Diabetes [hemoglobin A1c, (HbA1c) >7.5%].
* Severe or uncontrolled hypertension [resting Systolic Blood Pressure (SBP) >180 millimeters of mercury (mmHg), or resting Diastolic Blood Pressure (DBP) >110mmHg at screening period].
* Severe hypotension [resting SBP less than (<) 90mmHg, or resting DBP<50mmHg].
* Resting heart rate <60 beat per minute (bpm).
* Any contradiction to Bisoprolol according to label, including:
* Acute heart failure or during episodes of heart failure decompensation requiring intravenous inotropic therapy.
* Cardiogenic shock.
* Atrioventricular block of second or third degree (without a pacemaker).
* Sick sinus syndrome.
* Sinoatrial block.
* Slowed heart rate, causing symptoms (symptomatic bradycardia),
* Decreased blood pressure, causing symptoms (symptomatic hypotension),
* Severe bronchial asthma or severe chronic obstructive pulmonary disease.
* Sever forms of peripheral arterial occlusive disease and Raynaud's syndrome.
* Untreated phaeochromocytoma.
* Metabolic acidosis.
* Hypersensitivity to bisoprolol or to any of the excipients.
* Severe Arrhythmia including atrial fibrillation, atrial flutter, ventricular fibrillation, ventricular flutter or ventricular tachycardia.
* Significant valvular heart disease, congenital heart disease, pulmonary heart disease or perinatal heart disease.
* Acute pulmonary edema.
* Severe hepatic dysfunction, defined as:
* Serum Alanine Aminotransferase (ALT) > triple the upper limit of the normal range; and/or
* Serum Aspartate Aminotransferase (AST) > triple the upper limit of the normal value range and/or
* Severe renal dysfunction, defined as:
* Serum creatinine > twice the upper limit of the normal range
* Chronic Kidney Disease (glomerular filtration rate <45 Milliliter per minute).
* Hyperthyroidism or hypothyroidism.
* Severe infectious disease, example (eg) Human Immunodeficiency Virus positive or active tuberculosis.
* Severe autoimmune disease, e.g. lupus erythematosus, multiple sclerosis.
* Severe respiratory, digestive, hematological disease (including Anemia of Hb < 100 gram per litre) or tumor.
* Known to be hypersensitivity to Bisoprolol, or any of the excipient.
* Substance or alcohol abuse.
* Received heart transplantation or pacemaker implantation; revascularization treatment within 3 months; or plan to receive above treatment in 6 months.
* Currently undertaking other treatment that may affect the safety and/or efficacy evaluation, e.g. beta receptors agonists, et cetera.
* No legal ability or legal ability is limited.
* Subjects unlikely to cooperate in the study or with inability or unwillingness to give informed consent.
* Child-bearing period women without effective contraceptive measures, pregnancy and lactation.
* Participation in another clinical trial within the past 90 days.
* Other significant condition that in the Investigator's opinion would exclude the subject from the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-12-26 (Actual); Study Completion 2018-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono Co., Ltd., China
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences, Beijing, China

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bisoprolol
Started | 20
Completed | 0
Not Completed | 20
Not completed — Study termination | 20

BASELINE CHARACTERISTICS:
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.37 (13.931)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Resting Heart Rate at Week 6
Description: Heartbeats in each minute were calculated and averaged to obtain the resting heart rate.
Time Frame: Baseline, Week 6
Population: Data was not collected since the study was terminated early due to limited beta-blocker naive participants among newly diagnosed heart failure participants which led barrier to the recruitment.
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

2. Secondary Outcome: Change From Baseline in Resting Heart Rate at Week 3, 10 and 18
Description: Heartbeats in each minute were calculated and averaged to obtain the resting heart rate.
Time Frame: Baseline, Week 3, 10 and 18
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

3. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF) at Baseline, Week 14 and 26
Description: LVEF was defined as the fraction of blood (in percent) pumped out of the heart's left ventricular chamber with each heart beat and it is used to measure the cardiac output for the heart. Ultrasound cardiogram performed to measure LVEF.
Time Frame: Baseline, Week 14 and 26
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

4. Secondary Outcome: Left Ventricular End-Systolic Dimension (LVESD) at Baseline, Week 14 and 26
Description: Left Ventricular End-Systolic Dimension was measured by Ultrasound cardiogram.
Time Frame: Baseline, Week 14 and 26
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

5. Secondary Outcome: Left Ventricular End-diastolic Dimension (LVEDD) at Baseline, Week 14 and 26
Description: Left Ventricular End-diastolic Dimension was measured by Ultrasound cardiogram.
Time Frame: Baseline, Week 14 and 26
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

6. Secondary Outcome: Interventricular Septal Thickness (IVST) at Baseline, Week 14 and 26
Description: Interventricular septal thickness was measured by Ultrasound cardiogram.
Time Frame: Baseline, Week 14 and 26
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

7. Secondary Outcome: Ratio of Early (E) to Late (A) Ventricular Filling Velocities (E/A Ratio) at Baseline, Week 14 and Week 26
Description: Early to late ratio was measured by ultrasound cardiogram.
Time Frame: Baseline, Week 14 and Week 26
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants With Clinically Relevant Systolic and Diastolic Blood Pressure
Description: Blood pressure (systolic and diastolic) measurement was taken at sitting position, with the elbow at the same level with the heart. Number of participants with clinically relevant systolic and diastolic blood pressure reported based on the assessment of the investigator.
Time Frame: Screening (Week -2) up to Week 26
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Participants | 0

9. Secondary Outcome: Number of Participants With New York Heart Association (NYHA) Class
Description: The NYHA classification assesses the severity of symptoms of heart failure. Here NYHA class of II - IV was assessed. NYHA II: Slight limitation of physical activity, comfortable at rest, but ordinary physical activity results in undue breathlessness, fatigue or palpitation. NYHA III: Marked limitation of physical activity, comfortable at rest, but less than ordinary activity causes undue breathlessness, fatigue or palpitation. NYHA IV: Unable to carry on any physical activity without discomfort, symptoms at rest can be present. If any physical activity is undertaken, discomfort increased.
Time Frame: Baseline, Week 26
Population: The safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Participants
  Baseline: NYHA class II | 10
  Baseline: NYHA class III | 10
  Baseline: NYHA class IV | 0
  Week 26: NYHA class II | 2
  Week 26: NYHA class III | 1
  Week 26: NYHA class IV | 0
  Week 26: Not evaluated | 17

10. Secondary Outcome: Percentage of Participants With Resting Heart Rate Less Than 70 Beats Per Minute (Bpm) and More Than 55 Bpm
Description: Resting heart rate measurement was taken at sitting position for a continuous record of 3 minutes. Heartbeats in each minute was calculated and averaged to obtain the resting heart rate.
Time Frame: Baseline up to Week 26
Population: The safety population included all subjects who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
percentage of participants | 0

11. Secondary Outcome: Quality of Life Based on Minnesota Living With Heart Failure (MLHF) at Baseline and End of Treatment
Description: MLHF questionnaire has 21 items. Questions assess the impact of frequent physical symptoms of heart failure and the effects of heart failure on physical and social functions. Each question had a possible score of 0 (best) to 5 (worst), for a total of 0 to 105. The higher the summed score, the worse is the impact of heart failure on a participant's quality of life.
Time Frame: Baseline, end of treatment (Week 26)
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

12. Secondary Outcome: Quality of Life Based on the Medical Outcomes Study Item Short From Health Survey (SF-36) at Baseline and End of Treatment
Description: Short Form Health Survey (SF-36), an instrument composed by 8 subscales: Physical Functioning, Physical Role Function, Bodily Pain, General Health, Vitality, Social Functioning, Emotional Role Function and Mental Health. The individual question items (Likert scale 0-4) are first summed for each item under the various sections. Then, those summary scores are then standardized on a scale between 0 and 1 using the mean and standard deviation of the actual scores and finally, weighted to a scale between 0 and 100. The items contributing to a scale are scored so that a higher score represents better health, and they are averaged together to create the scale score. Each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively.
Time Frame: Baseline, end of treatment (Week 26)
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

13. Secondary Outcome: 6-Minute Walk Test
Description: 6-min walk test was a practical simple test that requires a 100-feet hallway but no exercise equipment or advanced training for technicians. Walking is an activity performed daily by all but the most severely impaired participants. This test measures the distance that a participant can quickly walk on a flat, hard surface in a period of 6 minutes.
Time Frame: Baseline and End of treatment (Week 26)
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Abnormal Value of N-terminal Pro-B-type Natriuretic Peptide (NT Pro-BNP)
Description: Routine blood tests was performed to measure NT Pro-BNP. The normal range for NT Pro-BNP varies from 0 picograms/milliliter (pg/mL) (lower limit of normal value) -125 pg/mL (upper limit of normal value).
Time Frame: Baseline up to End of treatment (Week 26)
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Participants | 19

15. Secondary Outcome: Mean 24 Hour, Day Time and Night Time Heart Rate
Description: Holter monitor was used to measure heart rate (24 hour, day time, night time).
Time Frame: Baseline, week 6, 14 and end of treatment (Week 26)
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Arrhythmia
Description: Holter monitor was used to diagnose arrhythmia.
Time Frame: Baseline up to end of treatment (Week 26)
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Participants | 0

17. Secondary Outcome: Number of Participants With 24 Hour Heart Rate With More Than 70 Beats Per Minute (Bpm) and Less Than 55 Bpm
Description: Holter monitor was used to measure heart rate.
Time Frame: Baseline, week 6, 14 and end of treatment (Week 26)
Population: The safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Participants | 0

18. Secondary Outcome: Number of Participants With Medicine Compliance Assessed by Medication Procession Ratio (MPR)
Description: MPR is used to assess the medicine compliance. MPR is defined as the actual drug number taken by the participants divided by the drug number should be taken by the participants according to the protocol. MPR between 80%-100% is defined as good compliance. Medication rate of less than (<) 80% or greater than (>)100% is defined as insufficient compliance.
Time Frame: Up to Week 26
Population: The safety population included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Participants
  MPR: Good Compliance | 18
  MPR: Insufficient compliance | 0
  Not evaluated | 2

19. Secondary Outcome: Number of Participants With All Cause Mortality, Cardiac Death, or Re-admission Due to Heart Failure
Description: Number of participants with all-cause mortality, cardiac death, or re-admission due to heart failure was reported.
Time Frame: Up to Week 26
Population: The safety population included all participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Bisoprolol
Number analyzed (Participants) | 20
Participants
  All-cause mortality | 1
  Cardiac death | 0
  Re-admission due to heart failure | 0

20. Primary Outcome: Change From Baseline in Resting Heart Rate at Week 14
Description: Heartbeats in each minute were calculated and averaged to obtain the resting heart rate.
Time Frame: Baseline, Week 14
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

21. Primary Outcome: Change From Baseline in Resting Heart Rate at Week 26
Description: Heartbeats in each minute were calculated and averaged to obtain the resting heart rate.
Time Frame: Baseline, Week 26
Population: as for outcome 1
Arm/Group | Bisoprolol
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Week 26
Arm/Group | Bisoprolol
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 4/20
Other Adverse Events (participants affected / at risk) | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=20)
Cardiac failure acute (Cardiac disorders) | 1
Sudden death (General disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bisoprolol (N=20)
Angina pectoris (Cardiac disorders) | 1
Sinoatrial block (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Upper respiratory tract infection 3 (15.0) (Infections and infestations) | 3
Blood uric acid increased (Investigations) | 1
Weight increased (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The study was terminated early due to limited beta-blocker naive participants among newly diagnosed heart failure participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03026088/Prot_SAP_000.pdf